CLINICAL TRIAL: NCT03042988
Title: Overnight Trials to Compare the Effects of Controlled Heat Stress Versus Sham Control on Nocturnal Supine Hypertension in Autonomic Failure Patients
Brief Title: Overnight Trials With Heat Stress in Autonomic Failure Patients With Supine Hypertension
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Italo Biaggioni, Professor of Medicine and Pharmacology, Vanderbilt University Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: VR22699; 141523 (Other: Vanderbilt IRB)
Record Dates: First submitted 2017-02-01; First posted 2017-02-03 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Hypertension; Pure Autonomic Failure; Multiple System Atrophy; Autonomic Failure
Keywords: supine hypertension; autonomic failure; heat stress; orthostatic hypotension
MeSH Terms: conditions — Hypertension; Pure Autonomic Failure; Multiple System Atrophy; Heat Stress Disorders; Hypotension, Orthostatic

STUDY DESIGN:
Intervention Model Description: randomized, 2-arm crossover study (heat vs sham)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Heat Stress (Experimental): Passive heat-stress using a commercial heating pad applied on the trunk
  Interventions: Other: Heating pad
- Control (Non-heating) (Sham Comparator): Commercial heating pad applied on the trunk but turned off
  Interventions: Other: Sham control

INTERVENTIONS:
Other: Heating pad — Heat stress applied on the trunk for up to 8 hours
  Other Names: Local heat stress
  Arms: Heat Stress
Other: Sham control — heating pad turned off applied on the trunk for up to 8 hours
  Other Names: control
  Arms: Control (Non-heating)

SUMMARY:
Patients with autonomic failure are characterized by disabling orthostatic hypotension (low blood pressure on standing), and at least half of them also have high blood pressure while lying down (supine hypertension). Exposure to heat, such as in hot environments, often worsens their orthostatic hypotension. The causes of this are not fully understood. The purpose of this study is to evaluate whether applying local heat over the abdomen of patients with autonomic failure and supine hypertension during the night would decrease their nocturnal high blood pressure while lying down. This will help us better understand the mechanisms underlying this phenomenon, and may be of use in the treatment of supine hypertension.

DETAILED DESCRIPTION:
Primary autonomic failure is a neurodegenerative condition characterized by loss of efferent sympathetic function and severe baroreflex impairment. The clinical hallmark of autonomic failure is disabling orthostatic hypotension, but at least half of patients are also hypertensive while lying down. This supine hypertension can be severe and associated with end-organ damage and worsening of orthostatic hypotension due to increased pressure natriuresis. It also complicates the management of these patients by limiting the use of daytime pressor agents for the treatment of orthostatic hypotension. Currently, no antihypertensive drug effectively lowers BP and prevents pressure natriuresis without worsening standing BP.

It is well known that heat exposure (e.g. hot weather or a hot bath or shower) produces an acute and temporary worsening of orthostatic hypotension in autonomic failure patients. Factors that may predispose these patients to the lowering BP effects of heat stress include 1) impaired heat dissipation due to inability to sweat, 2) preserved heat-mediated skin vasodilation, and 3) blunted sympathetic hemodynamic responses to maintain BP (increases in cardiac output, heart rate, and vaso- and venoconstriction). Our preliminary results showed that 2 hours of passive heat stress lowers BP in these patients through a decrease in central volume. In this study, we will assess the efficacy and safety of passive heat stress in the treatment of nocturnal supine hypertension in autonomic failure patients. Our hypothesis is that controlled local (abdominal) passive heat stress applied during the night will lower nocturnal BP in autonomic failure patients with supine hypertension.

To test this hypothesis, we propose to compare the BP effects of passive heat applied during the night vs. a sham control in a randomized crossover study in autonomic failure patients with supine hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients, between 18-80 yrs., with primary autonomic failure (Parkinson Disease, Multiple System Atrophy, and Pure Autonomic Failure) and supine hypertension. Supine hypertension will be defined as SBP≥150 mmHg.
* Patients able and willing to provide informed consent.

Exclusion Criteria:

* Pregnancy
* Significant cardiac, renal or hepatic illness, or with contraindications to administration of pressor agents or with other factors, which in the investigator's opinion would prevent the subject from completing the protocol including clinically significant abnormalities in clinical, mental or laboratory testing.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-01-30 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Systolic blood pressure | 10 pm - 8 am
  Maximal change from baseline in systolic blood pressure during the night, measured from 10 pm to 8 am

SECONDARY OUTCOMES:
Orthostatic Tolerance the following morning | 10 min standing
  Orthostatic tolerance defined as the area under the curve of standing systolic blood pressure calculated by the trapezoidal rule (upright systolic blood pressure multiplied by standing time) during a 10-minute standing test

CONTACTS AND LOCATIONS:
Overall Officials: Italo Biaggioni, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Autonomic Dysfunction Center/ Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Okamoto LE, Celedonio JE, Smith EC, Gamboa A, Shibao CA, Diedrich A, Paranjape SY, Black BK, Muldowney JAS 3rd, Peltier AC, Habermann R, Crandall CG, Biaggioni I. Local Passive Heat for the Treatment of Hypertension in Autonomic Failure. J Am Heart Assoc. 2021 Apr 6;10(7):e018979. doi: 10.1161/JAHA.120.018979. Epub 2021 Mar 19. PMID 33739123